CLINICAL TRIAL: NCT06602791
Title: The Effect of Watching Short Videos on Preoperative Anxiety in Pediatric Endoscopy Patients: A Prospective Randomized Study
Brief Title: The Effect of Watching Short Videos on Preoperative Anxiety
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, caner genc, Medical Doctor, Samsun University
Other Study IDs: Short videos in endoscopy
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Anesthesia; Anxiety
Keywords: anesthesia; anxiety; short videos; pediatric endoscopy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Video Group: Patients will be taken to the preoperative preparation unit, where those in the video group will watch short videos of their choice on a phone or tablet for 20 minutes under the guidance of their parents.
- Control Group (Standard): The control group will undergo standard preoperative preparation. Patients in this group will not watch any videos.

SUMMARY:
Preoperative anxiety is a common issue observed in pediatric patients prior to endoscopic procedures, and it can negatively affect the patient's overall experience. The aim of this study is to evaluate whether watching short videos on platforms such as YouTube Shorts, Instagram Reels, or TikTok has an impact on preoperative anxiety levels in pediatric endoscopy patients.

DETAILED DESCRIPTION:
The study was designed as a prospective randomized trial. Patients aged 6-12 years undergoing endoscopy and/or colonoscopy in the pediatric endoscopy unit will be divided into the video and the control groups. Patients will be taken to the preoperative preparation unit, where those in the video group will watch short videos of their choice on a phone/tablet for 20 minutes under the supervision of their parents. The control group will receive standard preoperative preparation. Anxiety levels will be assessed using the Modified Yale Preoperative Anxiety Scale (mYPAS) at six different time points: upon entry to the pre-procedural preparation room (T1), upon exiting the pre-procedural preparation room (T2), in the procedure room (T3), upon entry to the recovery unit (T4), at the 15th minute in the recovery unit (T5), and upon exiting the recovery unit (T6). Additionally, the indication for the procedure (e.g., celiac disease, Crohn's disease, ulcerative colitis), history of prior endoscopy/colonoscopy, oxygen saturation (SPO2%), heart rate (HR), mean arterial pressure (MAP) during the procedure, and the duration of monitoring in the recovery unit will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 5-12 years undergoing endoscopy and/or colonoscopy, classified as ASA I-II

Exclusion Criteria:

* Patients under 5, over 12, or with ASA score >2
* Epilepsy

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged 5-12 years undergoing endoscopy and/or colonoscopy, classified as ASA I-II will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Modified Yale Preoperative Anxiety Scale (mYPAS) scores | 1 hour
  Anxiety scores assessed and recorded at six distinct time points-namely, entry to the pre-procedural preparation room (T1), exit from the pre-procedural preparation room (T2), in the procedure room (T3), entry to the recovery unit (T4), at the 15th minute in the recovery unit (T5), and exit from the recovery unit (T6)-constitute the primary outcome of the study.

SECONDARY OUTCOMES:
Recovery Time | 1 hour
  The duration of patient monitoring in the recovery unit post-procedure, as assessed by the Modified Aldrete Score, is designated as the secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Caner Genc, M.D., Principal Investigator — Samsun University
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No